CLINICAL TRIAL: NCT05885204
Title: Robot-Assisted Versus Conventional Laparoscopic Radical Cystectomy in A Multicenter Cohort Study: A Propensity Score Matching Analysis
Brief Title: RARC vs LRC in A Multicenter Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-353-01
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Radical cystectomy; Robot-assisted laparoscopy; Conventional laparoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Sun Yat-sen Memorial Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- Renji Hospital, Shanghai Jiaotong University School of Medicine
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- The Third Medical Centre of Chinese PLA General Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- The First Affiliated Hospital of Nanchang University
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- Peking University Third Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- The Second Xiangya Hospital, Central South University
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- Zhongda Hospital Southeast University
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- The First Hospital of Jilin University
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- Second Hospital of Dalian Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy
- Gansu Provincial Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy; Procedure: Conventional laparoscopic radical cystectomy

INTERVENTIONS:
Procedure: Robot-assisted radical cystectomy — Robot-assisted laparoscopic radical cystectomy
Procedure: Conventional laparoscopic radical cystectomy — Conventional laparoscopic radical cystectomy

SUMMARY:
A multicenter, retrospective research was conducted. Patients who underwent robot-assisted radical cystectomy and laparoscopic radical cystectomy in 10 large medical centers in China were enrolled, comparing the oncologic outcomes of the patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old; Clinical stage Ta-T4a/N0-3/M0

Exclusion Criteria:

* Severe cardiovascular disease; History of previous major abdominopelvic surgery; Patients with distant metastases; Medical history of malignancy in other organs.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent robot-assisted radical cystectomy or laparoscopic radical cystectomy for bladder cancer from 2012 to 2021 in 10 large tertiary hospitals
Sampling Method: Probability Sample
Enrollment: 3815 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Five years
  Time from surgery until death from any cause.
Recurrence-free Survival | Five years
  Time from surgery to tumor recurrence which identified either pathologically or radiographically.
Cancer-specific Survival | Five years
  Time from date of surgery to death from bladder cancer.

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to privacy and ethical restrictions.